CLINICAL TRIAL: NCT07387003
Title: A Multicenter Phase 2 Clinical Study to Evaluate the Efficacy and Safety of GZR101-80 Injection in Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Oral Antidiabetic Drugs or Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Basal/Premixed Insulin
Brief Title: Evaluate the Efficacy and Safety of GZR101-80 Injection in Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR101-T2D-203
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR101-80 (Experimental)
  Interventions: Drug: GZR101-80
- Insulin degludec/Insulin aspart or Insulin aspart 30 (NovoRapid®30) (Active Comparator)
  Interventions: Drug: Insulin degludec/Insulin aspart or Insulin aspart30 (NovoRapid®30)

INTERVENTIONS:
Drug: GZR101-80 — Administered SC
  Arms: GZR101-80
Drug: Insulin degludec/Insulin aspart or Insulin aspart30 (NovoRapid®30) — Administered SC
  Arms: Insulin degludec/Insulin aspart or Insulin aspart 30 (NovoRapid®30)

SUMMARY:
This study will be conducted to evaluate the efficacy and safety of GZR101-80 Injection in patients with type 2 diabetes mellitus inadequately controlled on oral antidiabetic drugs or Basal/Premixed Insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects sign the Informed Consent Form (ICF) before the study, fully understand the contents, process and possible adverse reactions of the study, and are able to follow the contraindications and restrictions specified in this protocol.
2. At the age of 18-75 (inclusive) at the time of informed consent, male or female.
3. Body mass index (BMI) ≥18.5 and ≤35.0 kg/m2 at screening.
4. According to the diagnostic criteria and classification of diabetes mellitus issued by the World Health Organization (WHO) in 1999, and the supplementary diagnostic criteria recommended by WHO for diagnosis with Hemoglobin A1c (HbA1c) (2011), the time to diagnose T2DM is ≥ 180 days at screening.

Exclusion Criteria:

1. Confirmed or suspected type 1 diabetes mellitus or specific types of diabetes due to other causes (monogenic diabetes, cystic fibrosis, pancreatitis, drug- or chemical-induced diabetes, etc.) prior to screening.
2. Grade 3 hypoglycemia within 3 months before screening.
3. Subjects who have any diseases that may affect HbA1c testing at screening, or subjects who have donated blood, lost more than 400 mL of blood, or received blood transfusion within 3 months prior to screening.
4. Diagnosis of active malignant tumor within 5 years prior to screening (excluding adequately treated or resected non-metastatic basal or squamous cell skin cancer, in situ cancer of cervix, or prostate cancer in situ), or with a high suspicion of potential malignant tumor at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2027-04-22 (Estimated); Study Completion 2027-08-17 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) from baseline after 16 weeks of treatment. | Baseline , 16 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose (FPG) from baseline after 16 weeks of treatment | Baseline , 16 weeks
Safety Endpoints | Baseline , 17 weeks
  Number of adverse events (AEs) and serious adverse events (SAEs), and number and percent

CONTACTS AND LOCATIONS:
Locations (1):
- Gan & Lee Pharmaceuticals, Beijing, China